CLINICAL TRIAL: NCT06691152
Title: Efficacy and Safety Study of CD19 Universal CAR T Cells in Refractory Systemic Lupus Erythematosus
Brief Title: Efficacy and Safety of CD19 UCAR T Cells in Refractory Systemic Lupus Erythematosus
Acronym: SLE
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: The Children's Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Principal Investigator, Mao Jianhua, Principal Investigator, The Children's Hospital of Zhejiang University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PBC078
Record Dates: First submitted 2024-11-11; First posted 2024-11-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Systemic Lupus Erythematosus; CAR T-Cells; Pediatrics
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CAR T cell treatment group (Experimental): This trial was designed as an open, single-arm, multicenter, dose-increasing trial, three dose groups (1×10^7/kg, 3×10^7/kg, 6×10^7/kg) are set up, starting from the low dose group to explore the safe and effective dose.
  Interventions: Biological: CD19 Universal CAR-T cells

INTERVENTIONS:
Biological: CD19 Universal CAR-T cells — Three dose groups (1×10^7/kg, 3×10^7/kg, 6×10^7/kg) were set up, starting from the low dose group climbing to explore the safe and effective dose.

SUMMARY:
This is an investigator-initiated trial to evaluate the safety and efficacy of CD19 Universal CAR-T cells in the treatment of refractory systemic lupus erythematosus.

DETAILED DESCRIPTION:
Systemic lupus erythematosus (SLE) is a serious autoimmune disease that can lead to extensive damage in multiple organs and systems, ultimately resulting in disability and even death. Children with SLE are particularly at risk of organ damage, especially to the kidneys, and tend to have a more severe and protracted course of the disease compared to adults. Since 2019, CAR T-cell therapy has been successfully applied to autoimmune diseases. Clinical studies have demonstrated that targeted auto-CD19 CAR T-cells hold significant therapeutic potential for SLE. These cells effectively slow down the pathological progression of SLE and can also effectively treat severe cases. However, there are many limitations to the wide application of autologous CAR T-cells, autologous CAR T-cells are "personalized" products, which take a long time to produce, and their quality is affected by the patient's own physique, which is not conducive to scale and standardization. Besides, due to the personalized and complex preparation process of autologous CAR-T cell products, the costs are quite high which limits the promotion of use in the population. Compared with autologous CAR-T cell product, universal CAR-T cell products derived from healthy donors, it is not affected by the quantity and quality of the patient's T cells, leading to a high success rate in preparation. A single batch can meet the needs of hundreds of people, offering absolute advantages in time and cost. Compared to traditional autologous CAR-T cells, allogeneic universal CAR T-cells can greatly expand the accessibility of the product to patients, benefiting more patients. The purpose of this study is to assess the safety and efficacy of the CD19 universal CAR-T cells in the treatment of refractory SLE.

ELIGIBILITY:
Inclusion Criteria:

1. Age:≥5 years old;
2. Diagnosed with SLE according to the 2019 EULAR/ACR SLE classification criteria；Still in moderate to severe disease activity despite ≥3M of high dose glucocorticoids(prednisone≥1mg/kg/d or other equivalent amount of other steriod ), hydroxychloroquine and at least 2 of the following treatments(cyclophosphamide, MMF, azathioprine, methotrexate, cyclosporin, tacrolimus, sirolimus, leflunomide, telitacicept, Beliumab, and rituximab); or Intolerant to standard treatments;
3. SLEDAI 2K score≥8 points;
4. The functions of important organs are basically normal:

   Cardiac function: Left ventricular ejection fraction (LVEF) ≥55% with no obvious abnormality in electrocardiogram; Renal function: eGFR≥30ML/min/1.73m2； Liver function: Asparagus cochinchinensis transase (AST) and Alanine Aminotransferase (ALT)≤3.0 ULN, Total Bilirubin (TBIL) in serum ≤2.0×ULN; Lung function: No serious lung lesions, SpO2≥92%;
5. Met the standards of leukapheresis or intravenous blood collection, No contraindication for cell collection;
6. Negative pregnancy test for female Subjects of childbearing age, agree to take effective contraceptive measures the first year after CAR-T infusion;
7. Participants or their guardians agrees to participate in the clinical trial and sign the informed consent form which indicating that he/she understands the purpose and procedure of the clinical trial and is willing to participate in the study.

Exclusion Criteria:

1. Received CAR T cell therapy previously;
2. Central nervous system (CNS) disease: CNS neurolupus requires intervention within 60 days);
3. Active tuberculosis at the time of screening;
4. Have a history of congenital heart disease or acute myocardial infarction within 6 months prior to screening; Or severe arrhythmias (including multisource frequent supraventricular tachycardia, ventricular tachycardia, etc.); Or combined with moderate to massive pericardial effusion, serious myocarditis, etc; Or patients with unstable vital signs who need hypertensive drugs；
5. Suffer from other diseases that require long-term use of glucocorticoid or high-dose of immunosuppressive agents;
6. Uncontrollable infection, or active infection that requires systemic treatment within 1 week prior to screening；
7. History of organ transplantation or hematopoietic stem cell transplantation, or ≥Grade 2 GVHD within 2 weeks prior to screening；
8. Hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) positive and peripheral blood hepatitis B virus (HBV) DNA titer greater than the normal reference value range; Or hepatitis C virus (HCV) antibody positive and peripheral blood hepatitis C virus (HCV) RNA titer greater than the normal reference value range; Or positive for human immunodeficiency virus (HIV) antibodies; Or syphilis test positive; Or cytomegalovirus (CMV) DNA test positive;
9. Received live vaccine within 4 weeks before screening;
10. Tested positive in Blood pregnancy test；
11. Previous or concurrent malignancy；
12. Patients who participated in other clinical study within 3 months prior to enrollment;
13. Any other conditions that the investigators deem it unsuitable for the study.

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-10-30 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Adverse events related to CD19 universal CAR-T cells | 3 months
  Incidence and severity of AEs associated with CD19 universal CAR-T cells as assessed by CTCAE v5.0

SECONDARY OUTCOMES:
Proportion of patients achieving DORIS remission after CD19 universal CAR-T infusion | 6 months
  6M DORIS response rate
Proportion of patients achieving low disease activity status (LLDAS) after CD19 universal CAR-T infusion | 3 months and 6 months
  LLDAS maintenance rate at 3M and 6M
Proportion of patients achieving SRI-4 remission after CD19 universal CAR-T infusion | 3 months and 6 months
  SRI-4 response rate at 3M and 6M
Cellular kinetics | 6 months
  CAR transgene levels by quantitative polymerase chain reaction (qPCR) in peripheral blood.

CONTACTS AND LOCATIONS:
Overall Officials: Jianhua Mao, Principal Investigator — Children's Hospital, Zhejiang University School of Medicine
Locations (1):
- Children's Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mougiakakos D, Kronke G, Volkl S, Kretschmann S, Aigner M, Kharboutli S, Boltz S, Manger B, Mackensen A, Schett G. CD19-Targeted CAR T Cells in Refractory Systemic Lupus Erythematosus. N Engl J Med. 2021 Aug 5;385(6):567-569. doi: 10.1056/NEJMc2107725. No abstract available. PMID 34347960
- [Background] Muller F, Taubmann J, Bucci L, Wilhelm A, Bergmann C, Volkl S, Aigner M, Rothe T, Minopoulou I, Tur C, Knitza J, Kharboutli S, Kretschmann S, Vasova I, Spoerl S, Reimann H, Munoz L, Gerlach RG, Schafer S, Grieshaber-Bouyer R, Korganow AS, Farge-Bancel D, Mougiakakos D, Bozec A, Winkler T, Kronke G, Mackensen A, Schett G. CD19 CAR T-Cell Therapy in Autoimmune Disease - A Case Series with Follow-up. N Engl J Med. 2024 Feb 22;390(8):687-700. doi: 10.1056/NEJMoa2308917. PMID 38381673
- [Background] Charras A, Smith E, Hedrich CM. Systemic Lupus Erythematosus in Children and Young People. Curr Rheumatol Rep. 2021 Feb 10;23(3):20. doi: 10.1007/s11926-021-00985-0. PMID 33569643
- [Background] Neelapu SS, Tummala S, Kebriaei P, Wierda W, Gutierrez C, Locke FL, Komanduri KV, Lin Y, Jain N, Daver N, Westin J, Gulbis AM, Loghin ME, de Groot JF, Adkins S, Davis SE, Rezvani K, Hwu P, Shpall EJ. Chimeric antigen receptor T-cell therapy - assessment and management of toxicities. Nat Rev Clin Oncol. 2018 Jan;15(1):47-62. doi: 10.1038/nrclinonc.2017.148. Epub 2017 Sep 19. PMID 28925994